CLINICAL TRIAL: NCT02674880
Title: Use of High-molecular Weight Hyaluronan in Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Diseases Treated With Non-invasive Ventilation: Feasibility and Outcomes
Brief Title: Hyaluronic Acid in Acute Exacerbation of COPD - Duration Of Noninvasive Assistance
Acronym: HAEC-DONA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Raffaele Antonelli Incalzi, Professore Ordinario, Settore scientifico MED/09, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.1(15PT).15 ComEt-CBM; ES102605 (Other Grant/Funding Number: NIEHS grant number)
Record Dates: First submitted 2016-02-02; First posted 2016-02-05 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- HMW-HA (Experimental): HMW-HA (Yabro - 5 ml of saline containing 0.3% hyaluronic acid sodium salt) via nebulizer b.i.d.
  Interventions: Drug: HMW-HA
- Placebo (Placebo Comparator): 5 ml of saline via nebulizer b.i.d.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HMW-HA — Aerolized administration b.i.d.
  Other Names: Yabro
  Arms: HMW-HA
Other: Placebo — Standard therapy
  Arms: Placebo

SUMMARY:
The objective of this study is to test the effect of High Molecular Weight Hyaluronic Acid (HMW-HA) on Non Invasive Ventilation (NIV) effectiveness in patients admitted to a sub-intensive care unit for respiratory failure due to acute exacerbation of Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
The objective of this study is to test the effect of HMW-HA on NIV effectiveness in patients admitted to a sub-intensive care unit for respiratory failure due to acute exacerbation of COPD. The design is a parallel-arm, single-blind, placebo-controlled randomized clinical trial. Eighty patients, aged eighteen years or older, admitted for respiratory failure primarily due to COPD exacerbation and requiring non-invasive ventilation will be enrolled and randomized to the study treatment (active or placebo).

All patients will be treated with NIV delivered using a Hamilton C1 ventilator and medical therapy according to current guidelines (inhaled long-acting b2 agonists, inhaled long-acting anticholinergic, inhaled and systemic corticosteroids, antibiotics). Patients randomized to the active intervention group will also receive HMW-HA (Yabro® - 5 ml of saline containing 0.3% hyaluronic acid sodium salt) via nebulizer b.i.d., while patients randomized in the control group will receive a matching placebo. Patients will be treated until weaning or until NIV failure, defined as oro-tracheal intubation or death.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years of age or older
* Admitted for respiratory failure primarily due to COPD exacerbation
* Requiring non-invasive ventilation
* Respiratory distress, as evidenced by moderate-to-severe dyspnea and use of accessory muscles of respiration
* Hypercapnic respiratory failure
* High respiratory rate

Exclusion Criteria:

* Respiratory arrest or the need for immediate intubation
* Upper airways obstruction
* Facial trauma
* Inability to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Cumulative time on NIV | Day 1-10
  Cumulative duration of NIV in hours during the enrollement

SECONDARY OUTCOMES:
Rate of decline of time on NIV | Day 1-10
  rapidity of weaning from NIV

OTHER OUTCOMES:
Indices of NIV efficacy over one week of treatment | 7 days
  measures of effectiveness of ventilation in a week of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Antonelli Incalzi, MD, Principal Investigator — Università Campus Biomedico di Roma
Locations (1):
- Università Campus Biomedico di Roma, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galdi F, Pedone C, McGee CA, George M, Rice AB, Hussain SS, Vijaykumar K, Boitet ER, Tearney GJ, McGrath JA, Brown AR, Rowe SM, Incalzi RA, Garantziotis S. Inhaled high molecular weight hyaluronan ameliorates respiratory failure in acute COPD exacerbation: a pilot study. Respir Res. 2021 Feb 1;22(1):30. doi: 10.1186/s12931-020-01610-x. PMID 33517896